CLINICAL TRIAL: NCT05394168
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of HLX53 (an Anti-TIGIT Fc Fusion Protein) in Patients With Advanced/Metastatic Solid Tumors
Brief Title: A Phase I Clinical Study of HLX53 in Advanced/Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX53-FIH101
Record Dates: First submitted 2022-04-29; First posted 2022-05-27 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Advanced/Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX53 (Experimental): an anti-TIGIT Fc fusion protein
  Interventions: Biological: HLX53

INTERVENTIONS:
Biological: HLX53 — There are 5 preset dose groups, namely 30mg/QW, 150mg/QW, 400mg/QW, 1000mg/Q3W and 2000mg/Q3W, administered by intravenous infusion.

SUMMARY:
This phase I, first-in-human, open-label clinical study will evaluate the safety, tolerability, pharmacokinetic characteristics and preliminary efficacy of HLX53 (an anti-TIGIT Fc fusion protein) in patients with advanced/metastatic solid tumors.

DETAILED DESCRIPTION:
This study is an open-label phase I clinical study to evaluate the safety, tolerability , PK/PD and preliminary efficacy of HLX53 in patients with advanced/metastatic solid tumor. 11-30 subjects with advanced or metastatic solid tumors will be enrolled. The accelerated titration and traditional 3 + 3 dose escalation design will be implemented. Subjects will receive intravenous infusion of HLX53 at different doses according to the order of enrollment. There are 5 preset dose groups, namely 30mg/QW, 150mg/QW, 400mg/QW, 1000mg/Q3W and 2000mg/Q3W, administered by intravenous infusion. Observation period of DLT will last for 21 days after the first administration of HLX53. Maximum tolerated dose (MTD) definition: The highest dose level at which no more than 1 of 6 DLT-evaluable subjects developed DLT. At the MTD dose, at least 6 subjects were evaluable for DLT. When the MTD is determined, the MTD is usually used as the RP2D, or the RP2D is determined based on safety, PK/PD/ADA/NAb characteristics, and potential clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in clinical studies, full understanding of the trial, and signing of informed consent, willingness to follow and ability to complete the study in accordance with the requirements of the trial protocol.
* histologically or cytologically confirmed advanced/metastatic solid tumors or lymphoma, failure of standard therapy, or no standard therapy.
* Age ≥ 18 years and ≤ 75 years at the time of informed consent.
* Eastern Cooperative Oncology Group (ECOG) score 0 or 1.
* At least one measurable lesion according to RECISTv1.1 or 2014 Lugano (lymphoma) response evaluation criteria.
* Life expectancy of more than three months.
* Adequate hematological function.
* Adequate liver function.
* Adequate renal function
* Adequate cardiac function.
* Male and female subjects of childbearing potential must agree to use at least 1 highly effective method of contraception during the trial and for at least 6 months after the last dose of study drug.

Exclusion Criteria:

* Known history of serious allergy to the components of HLX53 or to any monoclonal antibody.
* Prior treatment with anti-TIGIT or antibody to the relevant target CD155, CD112, or CD113.
* Unresolved toxicity after prior antineoplastic therapy, i.e., not resolved to baseline, Grade 0-1 per NCI-CTCAE 5.0 (except alopecia).
* Coexisting unstable or controlled medical conditions.
* Spinal cord compression with clinical symptoms.
* Prior allogeneic bone marrow transplant or solid organ transplant.
* History of primary immunodeficiency.
* History of eczema or asthma that cannot be controlled by topical corticosteroids.
* History of any second malignancy within 2 years, except for curatively treated early malignancies (carcinoma in situ or stage I tumors) such as non-melanoma skin cancer, carcinoma in situ of the cervix, localized prostate cancer, ductal carcinoma in situ of the breast, papillary thyroid cancer.
* Vaccination with a live attenuated vaccine within 4 weeks prior to the first dos.e
* Use of immunosuppressive drugs within 2 weeks prior to initial administration.
* Received major surgery, anti-tumor therapy (chemotherapy, radiotherapy, targeted therapy, immunotherapy or biological therapy) within 4 weeks prior to the first dose.
* Known to have active infectious disease such as active HBV, HCV infection.
* History of human immunodeficiency virus (HIV) infection.
* Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-12-04 (Estimated); Study Completion 2025-03-04 (Estimated)

PRIMARY OUTCOMES:
Adverse event | Through study completion, assessed up to 2 years.
  Incidence and severity of adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 for patients receiving study drug.
Incidence of DLT | Up to 3 weeks.
  Ratio of the number of patients with DLT events in each dose group to the number of patients in the dose group during the DLT evaluation period.
MTD | Up to 3 weeks
  The maximum tolerated dose (MTD) of HLX53
RP2D | Through study completion, assessed up to 2 years.
  The recommended phase II dose (RP2D) of HLX53

SECONDARY OUTCOMES:
Cmax | From baseline to 30 days after the last administration, assessed up to 7 months
  Peak concentration of HLX53
Tmax | From baseline to 30 days after the last administration, assessed up to 7 months
  Time to reach peak concentration of HLX53
t1/2 | From baseline to 30 days after the last administration, assessed up to 7 months
  Elimination half-life of HLX53
TIGIT Receptor Occupancy | From baseline to 30 days after the last administration，assessed up to 7 months
  TIGIT Receptor Occupancy of HLX53 on Peripheral Circulating T Cells
ADA | From baseline to 30 days after the last administration，assessed up to 7 months
  Incidence of anti-drug antibodies (ADA)
Objective response rate (ORR) | Through study completion, assessed up to 2 years.
  Percentage of patients with complete response or partial response determined by investigators according to RECIST v1.1, iRECIST 2017 (solid tumors), or Lugano 2014 (lymphoma).
Progression-free survival (PFS) | From date of the first HLX53 administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years.
  PFS is defined as the time from the first administration of HLX53 to the first occurrence of disease progression or death due to any cause, whichever occurs first.
Overall survival(OS) | From date of the first HLX53 administration until the date of death from any cause, whichever came first, assessed up to 2 years.
  OS is defined as the time from the first administration of HLX53 to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China